CLINICAL TRIAL: NCT07285694
Title: An Open-label, Multicenter Phase 1/2 Study to Evaluate the Safety and Efficacy of AB-3028 in Patients With Castration Resistant Prostate Cancer (CRPC)
Brief Title: AB-3028, a Programmable Circuit T Cell Therapy in Patients With Castration Resistant Prostate Cancer (CRPC)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Arsenal Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AB-3028-201
Record Dates: First submitted 2025-12-10; First posted 2025-12-16 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Castration Resistant Prostate Cancer (mCRPC)
Keywords: prostate cancer; metastatic; Programmable circuit T cell; CRPC; AB-3028; autologous Cell Therapy; Cell Therapy; CAR T; castration resistant
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AB-3028 (Experimental): Patients receive a single dose of AB-3028 intravenously on day 0.
  Interventions: Biological: AB-3028

INTERVENTIONS:
Biological: AB-3028 — autologous T cell therapy

SUMMARY:
This is a multi-center, open-label Phase 1/2 trial evaluating the safety and efficacy of AB-3028 in subjects with metastatic castration resistant prostate cancer (mCRPC).

DETAILED DESCRIPTION:
This study is intended for subjects diagnosed with metastatic castration-resistant prostate cancer (mCRPC) and whose disease progressed after treatment with an androgen receptor pathway inhibitor (ARPI). The purpose of this study is to test the safety and efficacy of AB-3028 cells in subjects with metastatic castration-resistant prostate cancer. This treatment has not been approved by the Food and Drug Administration.

The goal of the Phase I portion of this study is to evaluate safety profile of AB-3028 and to determine the maximum tolerated dose or recommended phase 2 dose of AB-3028. The Phase 2 portion of the study will investigate the efficacy of AB-3028. T cells are part of the immune system that protect the body from infection and may help fight cancer. The T cells given in this study will come from the subject and will have a DNA cassette put in them that makes them able to recognize a priming antigen as well as Prostate-Specific Membrane Antigen (PSMA), two proteins found on prostate cancer tumor cells. These logic-gated T cells may help the body's immune system identify and kill cancer cells while sparing normal healthy tissues from toxicity.

The AB-3028 cells are given as a single intravenous infusion.

After completion of study treatment, subjects are followed with serial measurements of safety, tolerability and response.

This is a research study to obtain new information that may help people in the future.

ELIGIBILITY:
Key Inclusion Criteria:

1. At least 18 years of age at time of signing informed consent form.
2. Histologically confirmed adenocarcinoma of the prostate, meeting all of the following criteria:

   • Documented progressive metastatic castration-resistant prostate cancer (mCRPC) based on PCWG3 criteria.
3. Prior prostate cancer treatment with at least 1 novel androgen receptor pathway inhibitor (ARPI) therapy.

   • PSMA+ by PSMA PET.
   * Measurable disease by RECIST 1.1 criteria, or evaluable disease via measurable PSA (≥ 1 ng/mL) per PCWG3 criteria.
4. Adequate organ functions.

Key Exclusion Criteria:

1. Any prior systemic therapy for CRPC within 14 days prior to scheduled protocol required leukapheresis.
2. Central nervous system (CNS) metastatic disease, leptomeningeal disease, or cord compression.
3. Unwillingness to participate in an extended safety monitoring period.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 190 (Estimated)
Dates: Start 2026-01-09 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2031-05 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of AB-3028 | From AB-3028 infusion up to 24 months post-infusion
  To assess safety and tolerability of increasing dose levels of AB-3028 in successive cohorts of subjects with metastatic CRPC to determine the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) of AB-3028

OTHER OUTCOMES:
Phase 1 (Dose escalation and Backfill Cohorts): incidence of adverse events | From AB-3028 infusion up to 24 months post-infusion
  Defined as dose-limiting toxicities based on a Bayesian optimal interval (BOIN) design
Phase 2 (Cohort expansion): Objective response rate (ORR) | From AB-3028 infusion up to 24 months post-infusion
  ORR based on Independent Review Committee (IRC) assessment, defined as the proportion of subjects who have achieved a best overall response of CR or PR according to RECIST v1.1

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa and Holden Comprehensive Cancer Center, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No